CLINICAL TRIAL: NCT05234203
Title: The Impact of a Polyphenol-Rich Supplement on Epigenetic and Cellular Markers of Immune Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Big Bold Health, PBC (Industry)
Collaborators: TruDiagnostic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BBH-PRS-001
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Immunity Disorders; Aging; Inflammation
Keywords: Inflammaging; Immunosenescence; Polyphenol; Phytochemical; Phytonutrient; Tartary buckwheat; Fagopyrum tataricum
MeSH Terms: conditions — Immune System Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, single-arm, open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HTB Rejuvenate (Experimental): 4 capsules of study interventional supplement delivered as 2 capsules two times a day for 90 days.
  Interventions: Dietary Supplement: HTB Rejuvenate

INTERVENTIONS:
Dietary Supplement: HTB Rejuvenate — 90 days of BID dosing of 2 capsules of HTB Rejuvenate

SUMMARY:
This is a prospective, interventional, single-arm, open-label pilot study of 50 patients to evaluate the effect of a polyphenol-rich nutritional supplement on epigenetic and cellular markers of immune age.

DETAILED DESCRIPTION:
The objective of this study is to understand the impact of a polyphenol-rich supplement on measurements of epigenetic immune age and immune cell patterns germane to immune age over a 90-day period. The primary objective of this trial is to assess the effects of the supplement, HTB Rejuvenate™, on immune age markers. The secondary objective of this trial is to assess the effects of the supplement, HTB Rejuvenate, on leukocyte immune profiles including T cell subsets and granulocytes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnicity.
* Age Range - 18 - 85 (inclusive)
* Participant must be able to comply with treatment plan and laboratory tests including ability and willingness to perform home venous blood draw using Tasso device.
* Participant must be able to read, write and speak English fluently
* Participant must have an established primary care provider
* Participant must be willing and able to consume 4 capsules per day throughout the duration of study period

Exclusion Criteria:

* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Known immune system issues or immunodeficiency disease
* History of viral illness which could be reactivated by immune downregulation
* Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke) disease
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Participants infected with hepatitis C or HIV
* Body Mass Index (BMI) greater than or equal to 40 kilograms per meter squared
* Presence of active infection in previous 4 weeks
* Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the Clinical Investigator would render a participant unsuitable to participate in the study
* Unable or unwilling to provide required blood sample for testing
* Current or previous use of known prescription immunomodulating products (e.g. glucocorticoids, tumor necrosis factor (TNF)-alpha inhibitors) in the month prior to the start of the trial.
* Taking a concentrated polyphenol-focused supplement in the month prior to the start of the trial (e.g., quercetin, Epigallocatechin gallate (EGCG), resveratrol, curcumin, berberine, soy isoflavones, rutin, luteolin fisetin) or products that contain Tartary buckwheat
* A known history of blood dyscrasias including coagulopathy
* Current use of prescription anticoagulant medications
* Current pregnancy, planned attempts to conceive during study period or sexually active females not using contraception, as well as lactating/nursing females
* Current job that requires night-shift work
* Known allergy to polyphenolics
* Known allergy to buckwheat or Tartary buckwheat
* Investors or immediate family of investors in Big Bold Health
* Any person deemed by Clinical Investigator as low likelihood of complying with study protocol (e.g. evidence of history of non-compliance, history of poor follow-up, multiple or complex scheduling conflicts).
* Planned surgical procedure during study period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Epigenetic immune age | Change from baseline to 90 days
  Measurement of changes in methylation patterns on DNA related to immune age using the TruAge Biological Age test, which tests for methylation at 850,000 separate locations on DNA

SECONDARY OUTCOMES:
Leukocyte profiling | Change from baseline to 90 days
  Relative numbers of T cell subsets and granulocytes obtained using deconvolution analysis from epigenetic data obtained from the TruAge Biological Age test, which tests for methylation at 850,000 separate locations on DNA

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Bland, Ph.D, Principal Investigator — Big Bold Health; Austin D Perlmutter, MD, Study Director — Big Bold Health
Locations (1):
- Big Bold Health PBC, Bainbridge Island, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kontis V, Bennett JE, Mathers CD, Li G, Foreman K, Ezzati M. Future life expectancy in 35 industrialised countries: projections with a Bayesian model ensemble. Lancet. 2017 Apr 1;389(10076):1323-1335. doi: 10.1016/S0140-6736(16)32381-9. Epub 2017 Feb 22. PMID 28236464
- [Background] Gensous N, Garagnani P, Santoro A, Giuliani C, Ostan R, Fabbri C, Milazzo M, Gentilini D, di Blasio AM, Pietruszka B, Madej D, Bialecka-Debek A, Brzozowska A, Franceschi C, Bacalini MG. One-year Mediterranean diet promotes epigenetic rejuvenation with country- and sex-specific effects: a pilot study from the NU-AGE project. Geroscience. 2020 Apr;42(2):687-701. doi: 10.1007/s11357-019-00149-0. Epub 2020 Jan 24. PMID 31981007
- [Background] Fitzgerald KN, Hodges R, Hanes D, Stack E, Cheishvili D, Szyf M, Henkel J, Twedt MW, Giannopoulou D, Herdell J, Logan S, Bradley R. Potential reversal of epigenetic age using a diet and lifestyle intervention: a pilot randomized clinical trial. Aging (Albany NY). 2021 Apr 12;13(7):9419-9432. doi: 10.18632/aging.202913. Epub 2021 Apr 12. PMID 33844651
- [Background] Stojkovic L, Zec M, Zivkovic M, Bundalo M, Boskovic M, Glibetic M, Stankovic A. Polyphenol-Rich Aronia melanocarpa Juice Consumption Affects LINE-1 DNA Methylation in Peripheral Blood Leukocytes in Dyslipidemic Women. Front Nutr. 2021 Jun 17;8:689055. doi: 10.3389/fnut.2021.689055. eCollection 2021. PMID 34222308
- [Background] Sharma, R., & Padwad, Y. (2020). Perspectives of the potential implications of polyphenols in influencing the interrelationship between oxi-inflammatory stress, cellular senescence and immunosenescence during aging. Trends in Food Science & Technology, 98, 41-52. https://doi.org/10.1016/j.tifs.2020.02.004
- [Background] Santos JC, Ribeiro ML, Gambero A. The Impact of Polyphenols-Based Diet on the Inflammatory Profile in COVID-19 Elderly and Obese Patients. Front Physiol. 2021 Jan 12;11:612268. doi: 10.3389/fphys.2020.612268. eCollection 2020. PMID 33584335
- [Background] Bahramsoltani R, Ebrahimi F, Farzaei MH, Baratpourmoghaddam A, Ahmadi P, Rostamiasrabadi P, Rasouli Amirabadi AH, Rahimi R. Dietary polyphenols for atherosclerosis: A comprehensive review and future perspectives. Crit Rev Food Sci Nutr. 2019;59(1):114-132. doi: 10.1080/10408398.2017.1360244. Epub 2017 Sep 25. PMID 28812379
- [Background] Amiot MJ, Riva C, Vinet A. Effects of dietary polyphenols on metabolic syndrome features in humans: a systematic review. Obes Rev. 2016 Jul;17(7):573-86. doi: 10.1111/obr.12409. Epub 2016 Apr 15. PMID 27079631
- [Background] Sharma R, Padwad Y. Plant-polyphenols based second-generation synbiotics: Emerging concepts, challenges, and opportunities. Nutrition. 2020 Sep;77:110785. doi: 10.1016/j.nut.2020.110785. Epub 2020 Mar 2. PMID 32283341
- [Background] da Silveira Vasconcelos, M., de Oliveira, L. M. N., Mota, E. F., de Siqueira Oliveira, L., Gomes-Rochette, N. F., Nunes-Pinheiro, D. C. S., ... & de Melo, D. F. (2020). Consumption of rich/enrich phytonutrients food and their relationship with health status of population. In Phytonutrients in Food (pp. 67-101). Woodhead Publishing. https://doi.org/10.1016/B978-0-12-815354-3.00006-X
- [Background] Liu RH. Health benefits of fruit and vegetables are from additive and synergistic combinations of phytochemicals. Am J Clin Nutr. 2003 Sep;78(3 Suppl):517S-520S. doi: 10.1093/ajcn/78.3.517S. PMID 12936943
- [Background] Huda MN, Lu S, Jahan T, Ding M, Jha R, Zhang K, Zhang W, Georgiev MI, Park SU, Zhou M. Treasure from garden: Bioactive compounds of buckwheat. Food Chem. 2021 Jan 15;335:127653. doi: 10.1016/j.foodchem.2020.127653. Epub 2020 Jul 24. PMID 32739818
- [Background] Dziedzic K, Gorecka D, Szwengiel A, Sulewska H, Kreft I, Gujska E, Walkowiak J. The Content of Dietary Fibre and Polyphenols in Morphological Parts of Buckwheat (Fagopyrum tataricum). Plant Foods Hum Nutr. 2018 Mar;73(1):82-88. doi: 10.1007/s11130-018-0659-0. PMID 29435700
- [Background] Caputo M, Bona E, Leone I, Sama MT, Nuzzo A, Ferrero A, Aimaretti G, Marzullo P, Prodam F. Inositols and metabolic disorders: From farm to bedside. J Tradit Complement Med. 2020 Mar 24;10(3):252-259. doi: 10.1016/j.jtcme.2020.03.005. eCollection 2020 May. PMID 32670820
- [Background] Wieslander G, Fabjan N, Vogrincic M, Kreft I, Janson C, Spetz-Nystrom U, Vombergar B, Tagesson C, Leanderson P, Norback D. Eating buckwheat cookies is associated with the reduction in serum levels of myeloperoxidase and cholesterol: a double blind crossover study in day-care centre staffs. Tohoku J Exp Med. 2011 Oct;225(2):123-30. doi: 10.1620/tjem.225.123. PMID 21931228
- [Background] Nishimura, M., Ohkawara, T., Sato, Y., Satoh, H., Suzuki, T., Ishiguro, K., ... & Nishihira, J. (2016). Effectiveness of rutin-rich Tartary buckwheat (Fagopyrum tataricum Gaertn.)'Manten-Kirari'in body weight reduction related to its antioxidant properties: A randomised, double-blind, placebo-controlled study. Journal of Functional Foods, 26, 460-469. https://doi.org/10.1016/j.jff.2016.08.004
- [Background] Del Bo' C, Bernardi S, Marino M, Porrini M, Tucci M, Guglielmetti S, Cherubini A, Carrieri B, Kirkup B, Kroon P, Zamora-Ros R, Liberona NH, Andres-Lacueva C, Riso P. Systematic Review on Polyphenol Intake and Health Outcomes: Is there Sufficient Evidence to Define a Health-Promoting Polyphenol-Rich Dietary Pattern? Nutrients. 2019 Jun 16;11(6):1355. doi: 10.3390/nu11061355. PMID 31208133
- [Derived] Perlmutter A, Bland JS, Chandra A, Malani SS, Smith R, Mendez TL, Dwaraka VB. The impact of a polyphenol-rich supplement on epigenetic and cellular markers of immune age: a pilot clinical study. Front Nutr. 2024 Nov 18;11:1474597. doi: 10.3389/fnut.2024.1474597. eCollection 2024. PMID 39628466